CLINICAL TRIAL: NCT04232631
Title: Non-Invasive Testing to Evaluate Wound Healing in Diabetes
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Peter Crisologo, DPM, Professor, University of Texas Southwestern Medical Center
Other Study IDs: 2018-0386
Record Dates: First submitted 2019-07-12; First posted 2020-01-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- patients with diabetic foot ulcers: * Patient of the investigators
  * Diagnosis of diabetes mellitus
  * One or more moderate to severe diabetic foot ulcers/infections
  * 18-89 years of age
  Interventions: Device: SnapshotNIR, Kent Imaging
- Normal healthy volunteers: over 18 years of age have a foot
  Interventions: Device: SnapshotNIR, Kent Imaging

INTERVENTIONS:
Device: SnapshotNIR, Kent Imaging — Vascular imaging device

SUMMARY:
Normal group: We will collect normative data from healthy individuals to include baseline data, screening, and images. Up to 500 people will be enrolled and can include normal healthy volunteers, staff and students/trainees. Data will be collected one time with no follow up.

Patient group: We will prospectively collect data using one instrument (camera) (SnapshotNIR, Kent Imaging, Calgary, Alberta, Canada). We will collect non-contact imaging data before surgeries, during surgeries (if feasible), and during follow-up clinic visits. We will collect vascular data, demographic medical history, wound characteristics and measurements, frequency of debridement, off-loading, and clinic visits from existing medical records. We will collect lab data such as cultures glycosylated hemoglobin, hemoglobin and hematocrit, ESR, CRP and eGFR obtained per standard of care.

Imaging with this device is research-only.

DETAILED DESCRIPTION:
This is a prospective, observational study. All medical and surgical care provided to the patient group will be standard of care.

Patient group: Once a patient is identified as requiring vascular intervention or lower extremity ulceration (includes lower extremity wound of any cause, a surgical incision, a flap or graft) and consent to participation, their lower extremity will be imaged. They will be imaged preop, intraop (if feasible) and on post-op day 1 + or - 7 days if they require surgery and for each surgery related to the ulceration. They will also be imaged once a month in follow up for up to a total of 6 months or healing of the wound, determined by study physician.

Normal group: The normal group will have one-time imaging and data collection.

The Kent instrument does not touch the patient and is being evaluated to measure perfusion to predict wound healing, flap survival and amputation level healing. They are research only and not standard of care, and are not being used to determine care in the patient group.

ELIGIBILITY:
Investigator patients

Inclusion Criteria:

* Patient of the investigators
* Diagnosis of diabetes mellitus
* One or more moderate to severe diabetic foot ulcers/infections
* 18-89 years of age

Exclusion Criteria:

* Non-diabetic
* Is pregnant or plans to become pregnant
* Is nursing or actively lactating
* Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.
* Active alcohol or substance abuse in the opinion of the investigator that could impair the subject's ability to provide informed consent, participate in the study protocol or record study materials
* Patients with a history of poor compliance

Normal Healthy volunteers

Inclusion Criteria:

* Over 18
* Have a foot

Exclusion Criteria:

* Foot wounds
* Non-English speaking

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investgator's patients, normal healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluating the effectiveness of SnapshotNIR device to measure perfusion to predict wound healing, flap survival and amputation level healing. The device will report the oxygen saturation, oxyhemoglobin and deoxyhemoglobin levels in superficial tissue. | Three years
  To evaluate the effectiveness of the Kent instrument to measure perfusion to predict wound healing, flap survival and amputation level healing.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Crisologo, DPM, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No